CLINICAL TRIAL: NCT00856557
Title: Intervening to Prevent Contextual Errors in Medical Decision Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EDU 08-430
Record Dates: First submitted 2009-03-03; First posted 2009-03-05 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-10

CONDITIONS: Psychosocial Circumstances
Keywords: Patients with complex psychosocial needs

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Seminar and Practicum (Experimental): Seminar and practicum that occurs over 4 week period for internal medicine residents, designed to provide a systematic approach to identifying and addressing contextual factors essential to planning patient care.
  Interventions: Behavioral: Seminar and Practicum
- No intervention (No Intervention): No educational intervention.

INTERVENTIONS:
Behavioral: Seminar and Practicum — A 4 hour seminar and practicum for internal medicine residents designed to provide a systematic approach to identifying contextual factors essential to planning patient care.
  Arms: Seminar and Practicum

SUMMARY:
This study assessed whether a medical education intervention improves the quality of medical decision making in the care of patients with complex psychosocial -- or contextual -- needs that are essential to address when planning their care. A group of internal medicine residents were randomly assigned to participate in the seminar and practicum and then they, along with a control group that had not participated, were assessed for the quality of their clinical decision making and its impact on patient care. The study also assessed whether contextualization of care is associated with better patient health care outcomes

DETAILED DESCRIPTION:
We enrolled 139 internal medicine residents at 2 VA hospitals, Jesse Brown and Hines, in a randomized controlled design. Half participated in a 4 hour seminar series integrated into their ambulatory curriculum. Each month a total of 8 residents participated. Following the intervention there were 3 levels of assessment: (1) All participants, intervention and control, participated in a brief exercise interviewing 4 standardized patients (SPs). Note that we separately enlisted the assistance of 8 attending physicians to assist with case development for these SPs. (2) The research team subsequently enrolled 3 real patients from each physician's practice with "red flags" such as poor adherence, or missed visits, suggestive of contextual issues that need to be addressed. Physicians were scored on their performance at identifying the underlying contextual factors that account for these red flags and on formulating an appropriate plan of care. (3) The coders prospectively defined successful vs. unsuccessful outcomes for each case. At the follow up visit data was collected on whether the desired outcome was achieved. The analysis compared the skills, performance and outcomes of the intervention compared with the control group to determine the efficacy of training residents to individualize care.

ELIGIBILITY:
Inclusion Criteria:

* Internal Medicine Residency with continuity of care clinics at either Jesse Brown or Hines VA Medical Centers

Exclusion Criteria:

* All resident physicians who do not meet inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2009-10; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saul J. Weiner, MD, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (1):
- Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois, United States

REFERENCES:
- [Result] Weiner SJ, Kelly B, Ashley N, Binns-Calvey A, Sharma G, Schwartz A, Weaver FM. Content coding for contextualization of care: evaluating physician performance at patient-centered decision making. Med Decis Making. 2014 Jan;34(1):97-106. doi: 10.1177/0272989X13493146. Epub 2013 Jun 19. PMID 23784847
- [Result] Weiner SJ, Schwartz A, Sharma G, Binns-Calvey A, Ashley N, Kelly B, Dayal A, Patel S, Weaver FM, Harris I. Patient-centered decision making and health care outcomes: an observational study. Ann Intern Med. 2013 Apr 16;158(8):573-9. doi: 10.7326/0003-4819-158-8-201304160-00001. PMID 23588745
- [Result] Schwartz A, Weiner SJ, Harris IB, Binns-Calvey A. An educational intervention for contextualizing patient care and medical students' abilities to probe for contextual issues in simulated patients. JAMA. 2010 Sep 15;304(11):1191-7. doi: 10.1001/jama.2010.1297. PMID 20841532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Resident physicians were consented and recruited from two clinical training facilities on a rolling basis over 30 months.
Groups:
- Seminar and Practicum: Seminar and practicum that occurs over 4 week period for internal medicine residents, designed to provide a systematic approach to identifying and addressing contextual factors essential to planning patient care.
  Seminar and Practicum on Contextualizing Care: A 4 hour seminar and practicum for internal medicine residents designed to provide a systematic approach to identifying contextual factors essential to planning patient care.
Period: Overall Study
Arm/Group | Seminar and Practicum | No Intervention
Started | 62 | 76
Received Intervention/Control | 62 | 76
Tested With Standardized Patients | 62 | 76
With Patients With Contextual Flags | 50 | 60
Completed | 50 | 60
Not Completed | 12 | 16
Not completed — No patients with contextual flags | 12 | 16

BASELINE CHARACTERISTICS:
Population: Resident physicians in primary care.
Groups:
- Total: Total of all reporting groups
Arm/Group | Seminar and Practicum | No Intervention | Total
Number analyzed (Participants) | 62 | 76 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 76 | 138
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 43 | 74
  Male | 31 | 33 | 64
Region of Enrollment [Number; unit: participants]
  United States | 62 | 76 | 138
Year in residency [Number; unit: participants]
  Post Grad Yr (PGY) 1 | 7 | 12 | 19
  PGY2 | 31 | 45 | 76
  PGY3 | 24 | 19 | 43

OUTCOME MEASURES:

1. Primary Outcome: Health Outcome Improvement Rate
Description: A target health outcome improvement for each patient is prospectively defined at the first visit in which a contextual red flag is noted. The study outcome is what proportion of a physician's patients achieve their target health outcome improvement as documented in the medical record at 9 months post first visit.
Time Frame: After 9 months of the recorded visit
Measure: Mean (Standard Deviation); unit: proportion of physician's patients
Arm/Group | Seminar and Practicum | No Intervention
Number analyzed (Participants) | 50 | 60
proportion of physician's patients | 0.68 (0.37) | 0.59 (0.43)
Statistical Analysis 1: Comparison: Seminar and Practicum vs No Intervention; Null hypothesis is equal distribution of proportion of successful encounters among groups; Test type: Superiority or Other; p = 0.33, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Seminar and Practicum vs No Intervention; Considering all encounters (n=179) of all physicians for who outcomes were measured (n=111) together, are encounters in which physicians contextualized the plan of care more likely to be associated with target health outcome achievement than encounters in which physicians did not, controlling for clustering of encounters within physicians. (Generalized logistic mixed model, with random intercept for physician); Test type: Superiority or Other; p = .036, Mixed Models Analysis; Odds Ratio, log = 0.724, Standard Error of Mean 0.346

2. Secondary Outcome: Rate of Contextual Probing
Description: Proportion of encounters in which physician probed contextual red flags expressed by patients and identified via audio recordings.
Time Frame: During initial patient recordings
Measure: Mean (Standard Deviation); unit: proportion of physician's patients
Arm/Group | Seminar and Practicum | No Intervention
Number analyzed (Participants) | 62 | 76
proportion of physician's patients | .26 (.25) | .27 (.29)
Statistical Analysis 1: Comparison: Seminar and Practicum vs No Intervention; Test type: Superiority or Other; p = .99, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Rate of Contextual Planning
Description: Proportion of patient encounters in which the physician's plan of care addressed contextual factors identified in the audio recordings
Time Frame: During initial patient recordings
Measure: Mean (Standard Deviation); unit: proportion of physician's patients
Arm/Group | Seminar and Practicum | No Intervention
Number analyzed (Participants) | 62 | 76
proportion of physician's patients | .18 (.23) | .21 (.24)
Statistical Analysis 1: Comparison: Seminar and Practicum vs No Intervention; Test type: Superiority or Other; p = .39, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Groups:
- Seminar and Practium: Seminar and practicum that occurs over 4 week period for internal medicine residents, designed to provide a systematic approach to identifying and addressing contextual factors essential to planning patient care.
  Seminar and Practicum on Contextualizing Care: A 4 hour seminar and practicum for internal medicine residents designed to provide a systematic approach to identifying contextual factors essential to planning patient care.
Arm/Group | Seminar and Practium | No Intervention
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/76
Other Adverse Events (participants affected / at risk) | 0/62 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes